CLINICAL TRIAL: NCT05613153
Title: Peppermint Oil as an Alternative Treatment for Children With Bladder and Bowel Dysfunction: A Prospective Study
Brief Title: Peppermint Oil as a Treatment for Children With Bladder and Bowel Dysfunction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2206102
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Bladder and Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases | interventions — peppermint oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peppermint Oil (Experimental): Peppermint oil will be provided free of charge to participants under the trademark Pepogest produced by the maker Nature's Way® (dosage 0.2 mL, 181 mg peppermint oil).
  Interventions: Dietary Supplement: Peppermint Oil

INTERVENTIONS:
Dietary Supplement: Peppermint Oil — Participants weighing more than 40 kg will receive 2 peppermint oil capsules 3 times a day. Smaller children who weigh between 30 kg and 40 kg will receive 1 capsule of peppermint oil 3 times a day. All subjects will receive 8 weeks of treatment.

SUMMARY:
The goal of this clinical trial is to study the effect of peppermint oil in in children with bladder and bowel dysfunction.

The main question it aims to answer is: Does peppermint oil improve symptoms of bladder and bowel dysfunction among children?

Participants will:

* Be provided peppermint oil capsules to be taken 3 times daily for 8 weeks.
* At baseline and at a follow-up visit (8 weeks later), participants will be asked to complete the Vancouver Nonneurogenic Lower Urinary Tract Dysfunction/Dysfunctional Elimination Syndrome Questionnaire.

Researchers will compare baseline and follow-up questionnaire data for each participant to determine if there is improvement in symptoms of bladder and bowel dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-17 years and weighing 30kg or more with non-neurogenic bladder and bowel dysfunction who have failed behavioral therapy. Behavioral therapy, or also termed standard urotherapy, is defined as encompassing the following components [15]: Information and demystification; instruction on avoidance of holding maneuvers, regular bowel habits, proper voiding posture; lifestyle advice encompassing balanced fluid intake and diet, diminished caffeine, regular bladder and bowel emptying patterns; registration of symptoms and voiding habits with bladder diaries or frequency-volume charts; support and encouragement via regular follow up with caregiver. Failure of behavioral therapy is defined as no symptomatology improvement after adherence to behavioral therapy after 6 weeks.
* Participants must be able to swallow pills

Exclusion Criteria:

* Patients with neurogenic bladder, tethered cord, Society of Fetal Urology grade 3-4 hydronephrosis, vesicoureteral reflux, learning disabilities, or those who have undergone surgical therapy for bladder and bowel dysfunction will be excluded.
* Patients on medical therapy with oxybutynin within the last 30 days.
* Patients with hiatal hernia, severe gastrointestinal reflux or gallbladder disorders or on medications for these conditions will be excluded.
* Patient weighing less than 30 kg.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom score | 8 weeks
  Vancouver Nonneurogenic Lower Urinary Tract Dysfunction/Dysfunctional Elimination Syndrome Questionnaire Score. This includes 13 items scored using a 5-point Likert scale for each item. A score of 0 denotes no complaints and a score of 4 indicates severe symptoms. Range of scores 0-54, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi A. Stephany, MD, Principal Investigator — Children's Hospital, Orange County
Locations (1):
- Children's Hospital, Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaz GT, Vasconcelos MM, Oliveira EA, Ferreira AL, Magalhaes PG, Silva FM, Lima EM. Prevalence of lower urinary tract symptoms in school-age children. Pediatr Nephrol. 2012 Apr;27(4):597-603. doi: 10.1007/s00467-011-2028-1. Epub 2011 Oct 4. PMID 21969094
- [Background] Neveus T, von Gontard A, Hoebeke P, Hjalmas K, Bauer S, Bower W, Jorgensen TM, Rittig S, Walle JV, Yeung CK, Djurhuus JC. The standardization of terminology of lower urinary tract function in children and adolescents: report from the Standardisation Committee of the International Children's Continence Society. J Urol. 2006 Jul;176(1):314-24. doi: 10.1016/S0022-5347(06)00305-3. PMID 16753432
- [Background] Jiang R, Kelly MS, Routh JC. Assessment of pediatric bowel and bladder dysfunction: a critical appraisal of the literature. J Pediatr Urol. 2018 Dec;14(6):494-501. doi: 10.1016/j.jpurol.2018.08.010. Epub 2018 Aug 28. PMID 30297226
- [Background] Landgraf JM, Abidari J, Cilento BG Jr, Cooper CS, Schulman SL, Ortenberg J. Coping, commitment, and attitude: quantifying the everyday burden of enuresis on children and their families. Pediatrics. 2004 Feb;113(2):334-44. doi: 10.1542/peds.113.2.334. PMID 14754946
- [Background] Hagglof B, Andren O, Bergstrom E, Marklund L, Wendelius M. Self-esteem before and after treatment in children with nocturnal enuresis and urinary incontinence. Scand J Urol Nephrol Suppl. 1997;183:79-82. PMID 9165615
- [Background] Varlam DE, Dippell J. Non-neurogenic bladder and chronic renal insufficiency in childhood. Pediatr Nephrol. 1995 Feb;9(1):1-5. doi: 10.1007/BF00858952. PMID 7742205
- [Background] Bower WF, Yew SY, Sit KY, Yeung CK. Half-day urotherapy improves voiding parameters in children with dysfunctional emptying. Eur Urol. 2006 Mar;49(3):570-4. doi: 10.1016/j.eururo.2005.12.001. Epub 2006 Jan 4. PMID 16420968
- [Background] Arlen AM. Dysfunctional Voiders-Medication Versus Urotherapy? Curr Urol Rep. 2017 Feb;18(2):14. doi: 10.1007/s11934-017-0656-0. PMID 28213858
- [Background] Lazarus J. Intravesical oxybutynin in the pediatric neurogenic bladder. Nat Rev Urol. 2009 Dec;6(12):671-4. doi: 10.1038/nrurol.2009.214. Epub 2009 Nov 10. PMID 19901914
- [Background] Donnellan CA, Fook L, McDonald P, Playfer JR. Oxybutynin and cognitive dysfunction. BMJ. 1997 Nov 22;315(7119):1363-4. doi: 10.1136/bmj.315.7119.1363. No abstract available. PMID 9402781
- [Background] Ekhart C, Vries T, Hunsel FV. Psychiatric adverse drug reactions in the paediatric population. Arch Dis Child. 2020 Aug;105(8):749-755. doi: 10.1136/archdischild-2019-317933. Epub 2020 Feb 14. PMID 32060030
- [Background] Alammar N, Wang L, Saberi B, Nanavati J, Holtmann G, Shinohara RT, Mullin GE. The impact of peppermint oil on the irritable bowel syndrome: a meta-analysis of the pooled clinical data. BMC Complement Altern Med. 2019 Jan 17;19(1):21. doi: 10.1186/s12906-018-2409-0. PMID 30654773
- [Background] Kline RM, Kline JJ, Di Palma J, Barbero GJ. Enteric-coated, pH-dependent peppermint oil capsules for the treatment of irritable bowel syndrome in children. J Pediatr. 2001 Jan;138(1):125-8. doi: 10.1067/mpd.2001.109606. PMID 11148527
- [Background] Korterink JJ, Rutten JM, Venmans L, Benninga MA, Tabbers MM. Pharmacologic treatment in pediatric functional abdominal pain disorders: a systematic review. J Pediatr. 2015 Feb;166(2):424-31.e6. doi: 10.1016/j.jpeds.2014.09.067. Epub 2014 Nov 8. PMID 25449223
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Walle JV, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourol Urodyn. 2016 Apr;35(4):471-81. doi: 10.1002/nau.22751. Epub 2015 Mar 14. PMID 25772695
- [Background] Kligler B, Chaudhary S. Peppermint oil. Am Fam Physician. 2007 Apr 1;75(7):1027-30. PMID 17427617
- [Background] Chumpitazi BP, Kearns GL, Shulman RJ. Review article: the physiological effects and safety of peppermint oil and its efficacy in irritable bowel syndrome and other functional disorders. Aliment Pharmacol Ther. 2018 Mar;47(6):738-752. doi: 10.1111/apt.14519. Epub 2018 Jan 26. PMID 29372567
- [Background] Madisch A, Heydenreich CJ, Wieland V, Hufnagel R, Hotz J. Treatment of functional dyspepsia with a fixed peppermint oil and caraway oil combination preparation as compared to cisapride. A multicenter, reference-controlled double-blind equivalence study. Arzneimittelforschung. 1999 Nov;49(11):925-32. doi: 10.1055/s-0031-1300528. PMID 10604046
- [Background] Madisch A, Holtmann G, Mayr G, Vinson B, Hotz J. Treatment of functional dyspepsia with a herbal preparation. A double-blind, randomized, placebo-controlled, multicenter trial. Digestion. 2004;69(1):45-52. doi: 10.1159/000076546. Epub 2004 Jan 30. PMID 14755152
- [Background] May B, Kohler S, Schneider B. Efficacy and tolerability of a fixed combination of peppermint oil and caraway oil in patients suffering from functional dyspepsia. Aliment Pharmacol Ther. 2000 Dec;14(12):1671-7. doi: 10.1046/j.1365-2036.2000.00873.x. PMID 11121917
- [Background] Nash P, Gould SR, Bernardo DE. Peppermint oil does not relieve the pain of irritable bowel syndrome. Br J Clin Pract. 1986 Jul;40(7):292-3. No abstract available. PMID 3527248
- [Background] Afshar K, Mirbagheri A, Scott H, MacNeily AE. Development of a symptom score for dysfunctional elimination syndrome. J Urol. 2009 Oct;182(4 Suppl):1939-43. doi: 10.1016/j.juro.2009.03.009. Epub 2009 Aug 20. PMID 19695637
- [Background] Jafarov R, Ceyhan E, Kahraman O, Ceylan T, Dikmen ZG, Tekgul S, Dogan HS. Efficacy of transcutaneous posterior tibial nerve stimulation in children with functional voiding disorders. Neurourol Urodyn. 2021 Jan;40(1):404-411. doi: 10.1002/nau.24575. Epub 2020 Nov 18. PMID 33205852